CLINICAL TRIAL: NCT01443975
Title: Clinical Evaluation on the Use of the X-pander Device
Acronym: X-Pander
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Company Medichanical Engineering (Unknown)
Responsible Party: Sponsor
Other Study IDs: N-20110043
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthrosis; Total Hip Arthroplasty
Keywords: Total Hip Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Measurement with x-pander in acetabulum prior to inserting the artificial hip socket.
  Interventions: Procedure: x-pander

INTERVENTIONS:
Procedure: x-pander — Measurement of the size and quality of the bony acetabulum before mounting the artificial hip socket.

SUMMARY:
The purpose of this study is to clinically evaluate the use of the x-pander device.

DETAILED DESCRIPTION:
Clinical evaluation on the use of the x-pander device during THA-surgery

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for hip osteoarthrosis

Exclusion Criteria:

* Previous surgery of the actual hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients for primary THA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B. Laursen, MD, PhD, Principal Investigator — Orthopaedic Surgery Research Unit, Aalborg Hospital, Denmark
Locations (2):
- Denmark (2):
  - Ortopaedic Clinic, Farsoe Hospital, Aalborg University Hospital
  - Ortopaedic Clinic, Frederikshavn Hospital, Aalborg University Hospital